CLINICAL TRIAL: NCT06338540
Title: Relation of Caries Color to Caries Severity and Its Microbial Load in Primary Molars. A Clinical Study
Brief Title: Relation of Caries Color to Caries Severity and Its Microbial Load
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: A26020822
Record Dates: First submitted 2024-02-14; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2023-08

CONDITIONS: Relation of Caries Color
Keywords: Relation of Caries Color; History of pain; Caries severity; ICDAS; Microbial load; Radiograph

STUDY DESIGN:
Intervention Model Description: Group 1: Yellow caries color Group 2: dark brown caries color Group 3: light brown caries color Group 4: black caries color
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): Black caries color
  Interventions: Other: dark brown color of caries; Other: light brown color of caries; Other: yellow color of caries
- Group 2 (Experimental): Dark brown caries color
  Interventions: Other: Black color of caries; Other: light brown color of caries; Other: yellow color of caries
- Group 3 (Experimental): Light brown caries color
  Interventions: Other: Black color of caries; Other: dark brown color of caries; Other: yellow color of caries
- Group 4 (Experimental): Yellow caries color
  Interventions: Other: Black color of caries; Other: dark brown color of caries; Other: light brown color of caries

INTERVENTIONS:
Other: Black color of caries — observation of the dental caries color will be confirmed with standardized photographs illustrating , the black caries color related to history of pain , ICDAS , pulp exposed and microbial load
  Arms: Group 2; Group 3; Group 4
Other: dark brown color of caries — observation of the dental caries color will be confirmed with standardized photographs illustrating , the dark brown caries color related to history of pain , ICDAS , pulp exposed and microbial load
  Arms: Group 1; Group 3; Group 4
Other: light brown color of caries — observation of the dental caries color will be confirmed with standardized photographs illustrating , the light brown caries color related to history of pain , ICDAS , pulp exposed and microbial load
  Arms: Group 1; Group 2; Group 4
Other: yellow color of caries — observation of the dental caries color will be confirmed with standardized photographs illustrating , the yellow caries color related to history of pain , ICDAS , pulp exposed and microbial load
  Arms: Group 1; Group 2; Group 3

SUMMARY:
This study is to find the relation of caries color to caries severity and its microbial load in primary molars.

DETAILED DESCRIPTION:
This study is to investigate the relationship between the caries color to caries severity and its microbial load.

ELIGIBILITY:
Inclusion Criteria:

1. Their ages ranged from (4 to 7) years.
2. They were healthy, free from any chronic disease and had no previous anxiety disorder or medical disability such as the history of seizures or convulsion disorders, nystagmus, vertigo or equilibrium disorders, eye problems and autism.
3. Primary molars with class 1 caries, normal furcation and normal periapical bone structure
4. They were indicated for restorative treatment under local anesthesia.
5. They were not indicated for pharmacological management

Exclusion Criteria:

1. Primary molars with class 2 caries
2. Teeth with mobility
3. Periapical abscess
4. Fistula

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Caries color related to history of pain | Up to 12 weeks
  Four caries color ( black , dark brown , light brown , yellow ) related to history of pain ( no pain, positive elicited pain, spontaneous pain, and nocturnal pain )
Caries color related to ICDAS | Up to 12 weeks
  Four caries color ( black , dark brown , light brown , yellow ) related to ICDAS ( 3,4,5,6)
Caries color related to pulp exposed | Up to 12 weeks
  Four caries color ( black , dark brown , light brown , yellow ) related to pulp exposed ( pulp exposed , no pulp exposed)
Caries color related to microbial load | Up to 12 weeks
  Four caries color ( black , dark brown , light brown , yellow ) related to microbial load ( Streptococci mutans and Lactobacilli for caries biopsy )

CONTACTS AND LOCATIONS:
Overall Officials: Khaled A Habbal, Master, Principal Investigator — Researcher of Pediatric Dentistry , Faculty of Dentistry Mansoura University; Salwa M Awad, Prof, Study Director — Prof. of Pediatric Dentistry and Dental Public Health Faculty of Dentistry Mansoura University; Hossam E Hammouda, PhD, Study Director — Assistant Professor of Pediatric Dentistry Faculty of Dentistry Mansoura University
Locations (1):
- Mansoura university, Al Mansurah, Dakahlia Governorate, Egypt